CLINICAL TRIAL: NCT03131986
Title: Cessation of Tyrosine Kinase Inhibitors in Patients With Chronic-phase Chronic Myelogenous Leukaemia Who Achieve Stable Deep Molecular Response
Brief Title: Cessation of Tyrosine Kinase Inhibitors in Patients With Chronic-phase Chronic Myelogenous Leukaemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Prof Kwong Yok Lam, The University of Hong Kong
Other Study IDs: QMH-CML-001
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Leukemia, Myelogenous, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For analysis by cytogenetic/ molecular methods for better understanding of the disease biology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the debut of imatinib, the first tyrosine kinase inhibitor(TKI), more than two decades ago, the prognosis of patients with chronic myelogenous leukaemia (CML) has continued to improve. It has been shown that life expectancy of CML patients is approaching that of the general population nowadays. Currently, indefinite use of TKIs in patients with chronic-phase CML who achieve optimal response remains the standard practice. Nevertheless, the concepts of "treatment-free remission" and "functional" cure have been hotly discussed in recent years. A number of major international clinical trials have demonstrated that about 40-60% of CML patients who previously enjoyed deep molecular response on TKI manage to stay free from molecular relapse after cessation of TKI therapy.

Local experience of TKI cessation is lacking. This study aims to recruit patients diagnosed with CML, chronic phase who are treated with TKIs and remain in stable deep molecular response for at least two years. It is planned to stop TKI in these patients with regular monitoring, and determine their outcomes.

DETAILED DESCRIPTION:
Major clinical trials including multicentre Stop Imatinib (STIM) trial, According to Stop Imatinib (A-STIM), TWISTER, Korean Imatinib Discontinuation Study (KIDS), European Stop Tyrosine Kinase Inhibitor Trial (EURO-SKI), and stop second generation (2G-TKI) showed that it is safe to stop TKI in patients who achieve stable deep molecular response (DMR) as defined by respective study groups. Around 40-60% of study participants managed to remain in treatment-free remission (TFR). For patients who experience molecular relapse after TKI withdrawal, most do so within the first 6 months. In addition, they all remained sensitive to TKI and majority of them were able to achieve the original molecular response. No loss of complete haematological response or progression to advanced phase CML was observed when the TKI was stopped.

Cessation of TKI in selected CML patients leads to freedom from treatment-related toxic effects. It is expected that at least 40% of enrolled patients will be in a sustained molecular remission after stopping TKI. Successful cessation would also reduce long-term treatment costs.

After cessation of TKI, fluctuation in molecular response, or even molecular relapse of the disease might bring about anxiety and distress in the patients. Some patients, estimated at around 40-60%, would experience molecular relapse and require resumption of TKI. Close molecular monitoring real-time polymerase chain reaction (RT-QPCR) after stopping TKI (every month in the first year and every 2 months in the second year) will allow early detection of possible molecular relapse and thus prompt resumption of TKI. Long-term risks of disease progression and drug resistance are uncertain, though the safety data from the TFR studies reported to date are sufficiently reassuring. Some patients might have musculoskeletal pain and pruritus after cessation of TKI, especially imatinib, which is also commonly known as "imatinib withdrawal syndrome".

Patients with chronic-phase CML who have been treated with a tyrosine kinase inhibitor for more than 3 years and had deep molecular response (breakpoint cluster region/Abelson murine leukemia (BCR-ABL1) transcript ≤0.0032% IS ratio, i.e. molecular response (MR4.5) for at least 2 years

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 years or above) patients diagnosed with chronic-phase CML
* In deep molecular response (i.e. MR4.5 or below, or those whose breakpoint cluster region -Abelson murine leukemia (BCR-ABL) transcripts were undetectable with at least 20,000 amplified copies of the control gene) for at least 2 years, confirmed by at least 3 data points with no more than one assessment between MR4 and MR4.5
* Under treatment with a TKI in first line, or in second line due to intolerance of another first-line TKI
* At least three years of treatment with the same TKI before enrolment

Exclusion Criteria:

* Under 18 years old
* Adults under law protection or without ability to consent
* Previous or planned autologous/allogeneic haematopoietic stem cell transplantation
* Documented kinase domain mutation
* History of disease progression (accelerated or blast phase)
* A change to the current TKI because of unsatisfactory response to a previous TKI in those who are on second line TKI (Note: patients are still considered eligible if the switch of TKI was due to intolerance or side effects)
* Patients who can speak neither Chinese nor English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients on TKI treatment for at least 3 years and DMR for at least 24 months and potentially eligible for the study will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 12 months
  molecular relapse-free survival without treatment

SECONDARY OUTCOMES:
disease free survival | 24 months
  molecular relapse-free survival without treatment
Overall survival | 24 months
  Overall survival without treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuk Man Cheung, MBBS(HK), Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Result] Rousselot P, Charbonnier A, Cony-Makhoul P, Agape P, Nicolini FE, Varet B, Gardembas M, Etienne G, Rea D, Roy L, Escoffre-Barbe M, Guerci-Bresler A, Tulliez M, Prost S, Spentchian M, Cayuela JM, Reiffers J, Chomel JC, Turhan A, Guilhot J, Guilhot F, Mahon FX. Loss of major molecular response as a trigger for restarting tyrosine kinase inhibitor therapy in patients with chronic-phase chronic myelogenous leukemia who have stopped imatinib after durable undetectable disease. J Clin Oncol. 2014 Feb 10;32(5):424-30. doi: 10.1200/JCO.2012.48.5797. Epub 2013 Dec 9. PMID 24323036
- [Result] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Yeung DT, Dang P, Goyne JM, Slader C, Filshie RJ, Mills AK, Melo JV, White DL, Grigg AP, Hughes TP. Safety and efficacy of imatinib cessation for CML patients with stable undetectable minimal residual disease: results from the TWISTER study. Blood. 2013 Jul 25;122(4):515-22. doi: 10.1182/blood-2013-02-483750. Epub 2013 May 23. PMID 23704092
- [Result] Lee SE, Choi SY, Song HY, Kim SH, Choi MY, Park JS, Kim HJ, Kim SH, Zang DY, Oh S, Kim H, Do YR, Kwak JY, Kim JA, Kim DY, Mun YC, Lee WS, Chang MH, Park J, Kwon JH, Kim DW. Imatinib withdrawal syndrome and longer duration of imatinib have a close association with a lower molecular relapse after treatment discontinuation: the KID study. Haematologica. 2016 Jun;101(6):717-23. doi: 10.3324/haematol.2015.139899. Epub 2016 Feb 17. PMID 26888022